CLINICAL TRIAL: NCT06603077
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of AVTX-009 in Patients With Moderate to Severe Hidradenitis Suppurativa (LOTUS)
Brief Title: A Study to Evaluate the Efficacy and Safety of AVTX-009 in Patients With Moderate to Severe Hidradenitis Suppurativa
Acronym: LOTUS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVTX-009-HS-201
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; HS; acne inversa; AVTX-009; LY2189102; FL-101
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AVTX-009 Regimen 1 (Experimental): Patients will receive AVTX-009 regimen 1.
  Interventions: Drug: AVTX-009 Regimen 1
- AVTX-009 Regimen 2 (Experimental): Patients will receive AVTX-009 regimen 2.
  Interventions: Drug: AVTX-009 Regimen 2
- Placebo (Placebo Comparator): Patients will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVTX-009 Regimen 1 — AVTX-009 will be administered as a subcutaneous injection every 4 weeks.
  Arms: AVTX-009 Regimen 1
Drug: AVTX-009 Regimen 2 — AVTX-009 will be administered as a subcutaneous injection every 2 weeks.
  Arms: AVTX-009 Regimen 2
Drug: Placebo — Matching placebo will be administered as a subcutaneous injection every 2 weeks.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of AVTX-009 compared with placebo in patients with moderate to severe Hidradenitis Suppurativa (HS).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, Phase 2 study. Patients will be randomized to one of two AVTX-009 dose regimens or matching placebo in a 1:1:1 ratio.

The study will comprise:

1. A Screening Period which will last up to 28 days.
2. A Treatment Period up to 16 weeks.
3. A Follow-up period of 6 weeks after the last dose of study drug.

The maximum clinical trial duration for each participant is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of hidradenitis suppurativa (HS) for at least 6 months prior to Screening.
2. At least 5 inflammatory lesions in at least 2 distinct anatomical areas, at least 1 of which is Hurley Stage 2 or 3.

Exclusion Criteria:

1. Has a draining fistula count of ≥ 20.
2. Has another active skin inflammatory condition, infection (viral, bacterial, or fungal), or another active ongoing inflammatory disease (other than HS) that requires treatment with a prohibited medication, which could interfere with the assessment of HS.
3. History of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic lung infection, recurrent urinary tract infection, or open, draining or infected skin wounds or ulcers (not related to HS).
4. Has severe, progressive and/or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or immunosuppressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | At Week 16
  HiSCR75 is defined as at least a 75% reduction in the total abscess and inflammatory nodule count, with no increase in abscess count and no increase in draining fistula count, relative to Baseline.

SECONDARY OUTCOMES:
Proportion of patients achieving HiSCR50 | At Week 16
  HiSCR50 is defined as at least a 50% reduction in the total abscess and inflammatory nodule count, with no increase in abscess count and no increase in draining fistula count, relative to Baseline.
Proportion of patients achieving HiSCR90 | At Week 16
  HiSCR90 is defined as at least a 90% reduction in the total abscess and inflammatory nodule count, with no increase in abscess count and no increase in draining fistula count, relative to Baseline.
Change from Baseline in International HS Severity Score System (IHS4) | Baseline (Day 1) and Week 16
  IHS4 score is calculated by the number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild disease, 4 to 10 signifies moderate disease, and 11 or higher signifies severe disease.
Change from Baseline in total abscess and inflammatory nodule (AN) count | Baseline (Day 1) and Week 16
  An abscess is a circumscribed collection of purulent exudates frequently associated with swelling, erythema, and other signs of inflammation, such as fluctuance, tenderness, and pain. An inflammatory nodule is a raised, deep-seated, three-dimensional, round nodule, greater than 10 mm in diameter. It is tender and erythematous without evidence of fluctuance.
Change from Baseline in draining fistula count | Baseline (Day 1) and Week 16
  Draining fistula is defined as a pathologic passageway connecting to the skin surface from dermis or subcutaneous tissue that drains serous or purulent fluid, either spontaneously or by gentle palpation.
Percentage of patients achieving at least a 30% reduction and at least a 1-unit reduction from Baseline on a Numerical Rating Scale (NRS) in Patient's Global Assessment of Skin Pain (PGA Skin Pain) among subjects with Baseline NRS ≥3 (NRS30) | Baseline (Day 1) and Week 16
  The skin pain NRS is a single-item measure to capture the patient's self-reported skin pain severity by rating the worst level of skin pain in the last 24 hours as a number on a numerical rating scale from 0 (no pain) to 10 (worst pain imaginable).
Percentage of patients with flares | From Baseline (Day 1) to Week 16
  The number of patients with flares will be programmatically calculated based on the assessed lesion counts. A flare is defined as ≥ 25% increase in AN count plus an increase of ≥ 2 in AN count compared to Baseline.
AVTX-009 anti-drug antibodies (ADA) | From Baseline (Day 1) to Week 20
  The incidence of patients with AVTX-009 anti-drug antibodies (ADA).
Safety and tolerability of AVTX-009 | From Baseline (Day 1) to Week 20
  Incidence of adverse events (AEs).

CONTACTS AND LOCATIONS:
Locations (89):
- United States (36):
  - Clinical Site 1022, Scottsdale, Arizona
  - Clinical Site 1037, Scottsdale, Arizona
  - Clinical Site 1026, Tucson, Arizona
  - Clinical Site 1032, Northridge, California
  - Clinical Site 1019, Pomona, California
  - Clinical Site 1009, Sacramento, California
  - Clinical Site 1034, Santa Monica, California
  - Clinical Site 1011, Washington D.C., District of Columbia
  - Clinical Site 1029, Boca Raton, Florida
  - Clinical Site 1002, Coral Gables, Florida
  - Clinical Site 1015, Maitland, Florida
  - Clinical Site 1027, North Miami Beach, Florida
  - Clinical Site 1013, Tampa, Florida
  - Clinical Site 1008, Savannah, Georgia
  - Clinical Site 1014, Chicago, Illinois
  - Clinical Site 1028, West Lafayette, Indiana
  - Clinical Site 1031, Bowling Green, Kentucky
  - Clinical Site 1024, Murray, Kentucky
  - Clinical Site 1042, Boston, Massachusetts
  - Clinical Site 1001, Boston, Massachusetts
  - Clinical Site 1030, Detroit, Michigan
  - Clinical Site 1007, Fort Gratiot, Michigan
  - Clinical Site 1041, Oakland, Michigan
  - Clinical Site 1003, Portsmouth, New Hampshire
  - Clinical Site 1036, Brooklyn, New York
  - Clinical Site 1016, New York, New York
  - Clinical Site 1023, The Bronx, New York
  - Clinical Site 1020, Cincinnati, Ohio
  - Clinical Site 1010, Cleveland, Ohio
  - Clinical Site 1017, Dublin, Ohio
  - Clinical Site 1004, Philadelphia, Pennsylvania
  - Clinical Site 1035, Pittsburgh, Pennsylvania
  - Clinical Site 1018, Johnston, Rhode Island
  - Clinical Site 1025, Providence, Rhode Island
  - Clinical Site 1005, Greenville, South Carolina
  - Clinical Site 1012, Arlington, Texas
- Australia (4):
  - Clinical Site 1203, Darlinghurst, New South Wales
  - Clinical Site 1201, Westmead, New South Wales
  - Clinical Site 1204, Woolloongabba, Queensland
  - Clinical Site 1202, Carlton, Victoria
- Bulgaria (4):
  - Clinical Site 1303, Sofia, Sofia-Grad
  - Clinical Site 1302, Lovech
  - Clinical Site 1301, Pleven
  - Clinical Site 1304, Stara Zagora
- Canada (9):
  - Clinical Site 1105, Edmonton, Alberta
  - Clinical Site 1108, Edmonton, Alberta
  - Clinical Site 1103, Barrie, Ontario
  - Clinical Site 1104, Hamilton, Ontario
  - Clinical Site 1107, London, Ontario
  - Clinical Site 1106, Toronto, Ontario
  - Clinical Site 1110, Montreal, Quebec
  - Clinical Site 1101, Saskatoon, Saskatchewan
  - Clinical Site 1111, Québec
- Czechia (2):
  - Clinical Site 1401, Prague, Prague
  - Clinical Site 1402, Prague, Prague
- France (5):
  - Clinical Site 1503, Antony, Hauts-de-Seine
  - Clinical Site 1505, Amiens, Picardie
  - Clinical Site 1502, Lyon, Rhône
  - Clinical Site 1501, Rouen, Seine-Maritime
  - Clinical Site 1504, Paris, Île-de-France Region
- Germany (5):
  - Clinical Site 1606, Erlangen, Bavaria
  - Clinical Site 1604, Frankfurt am Main, Hesse
  - Clinical Site 1601, Bochum, North Rhine-Westphalia
  - Clinical Site 1602, Münster, North Rhine-Westphalia
  - Clinical Site 1605, Dresden, Saxony
- Greece (3):
  - Clinical Site 2103, Athens, Attica
  - Clinical Site 2101, Athens, Attica
  - Clinical Site 2102, Efkarpia, Thessaloniki
- Italy (7):
  - Clinical Site 1901, Torrette, Ancona
  - Clinical Site 1903, Rozzano, Milano
  - Clinical Site 1902, Ferrara
  - Clinical Site 1908, Milan
  - Clinical Site 1906, Pisa
  - Clinical Site 1907, Roma
  - Clinical Site 1904, Roma
- Poland (6):
  - Clinical Site 1702, Wroclaw, Kuyavian-Pomeranian Voivodeship
  - Clinical Site 1706, Wroclaw, Lower Silesian Voivodeship
  - Clinical Site 1703, Bialystok, Podlaskie Voivodeship
  - Clinical Site 1701, Warszawa, Pomeranian Voivodeship
  - Clinical Site 1705, Warszawa, Pomeranian Voivodeship
  - Clinical Site 1704, Ossy, Silesian Voivodeship
- Slovakia (2):
  - Clinical Site 2202, Svidník, Presov
  - Clinical Site 2201, Trnava, Trnava Region
- Spain (4):
  - Clinical Site 1801, Manises, Valencia
  - Clinical Site 1802, Granada
  - Clinical Site 1803, Madrid
  - Clinical Site 1804, Seville
- Turkey (Türkiye) (2):
  - Clinical Site 2001, Gaziantep
  - Clinical Site 2002, Samsun

IPD SHARING:
Plan to Share IPD: No